CLINICAL TRIAL: NCT04539197
Title: Detection of Circulating Plasmablast in Diagnosis and Relapse Prediction of IgG4 Related Diseases
Brief Title: Circulating Plasmablast in Diagnosis and Relapse Prediction of IgG4-RD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Plasmablast in IgG4-RD
Record Dates: First submitted 2020-09-01; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-06

CONDITIONS: Plasmablast/Plasma Cells in Diagnosis of IgG4-RD; Plasmablast/Plasma Cells in Relapse Prediction of IgG4-RD
Keywords: IgG4 related disease; plasmablast/plasma cells; diagnosis; relapse
MeSH Terms: conditions — Immunoglobulin G4-Related Disease; Disease; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — 3-5 ml peripheral blood was collected for PBMC seperation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- IgG4-RD group: 300 IgG4-RD were enrolled and followed up for more than 6 months. Peripheral blood of all patients were collected at baseline, disease remission and relpase for plasmablast/plasma cells detection. All clinical data and laboratory parameters at baseline, each follow up were collected.
- other autoimmune disease group: 200 patients( RA, SLE, pSS, BD, et al) were enrolled in this study. Peripheral blood of all patients were collected at baseline for plasmablast/plasma cells detection. All clinical data and laboratory parameters at baseline were collected.
- IgG4-RD mimicker group: 60 IgG4-RD mimickers (pancreatic cancer, cholangiocarcinoma, vasculitis, lymphoproliferative diseases, inflammatory bowel disease, kimura disease) were collected. Peripheral blood of all patients were collected at baseline for plasmablast/plasma cells detection. All clinical data and laboratory parameters at baseline were collected.
- healthy control group: 100 healthy controls were collected. Peripheral blood of healthy controls were collected at baseline for plasmablast/plasma cells detection. Demographic features of healthy controls were collected.

SUMMARY:
300 IgG4-RD patients, 200 other autoimmune diseases, 60 IgG4-RD mimickers and 100 healthy controls were enrolled. Circulating plasmablast/plasma cells were detected of all patients at baseline and healthy controls. IgG4-RD patients were followed up every 3-6 months. Circulating plasmablast/plasma cells were also detected at disease remission and relapse. IgG4-RD patients' clinical data and laboratory parameters were collected.

DETAILED DESCRIPTION:
300 IgG4-RD patients, 200 other autoimmune diseases, 60 IgG4-RD mimickers (pancreatic cancer, cholangiocarcinoma, vasculitis, lymphoproliferative diseases, inflammatory bowel disease, kimura disease) and 100 healthy controls were enrolled. Peripheral blood samples of 5-10 ml were collected from all patients and healthy controls. Serum was separated for ELISA detection. Circulating plasmablast/plasma cells were detected of all patients at baseline and healthy controls. IgG4-RD patients were followed up every 3-6 months. Circulating plasmablast/plasma cells were also detected at disease remission and relapse. IgG4-RD patients' clinical data and laboratory parameters were collected. Data were analyzed to evaluate plasmablast/plasma cells in diagnosis and relapse prediction of IgG4-RD.

ELIGIBILITY:
Inclusion Criteria:

* IgG4-RD patients fulfilled the 2011 comprehensive diagnostic criteria of IgG4-RD (2011). Other autoimmune disease and IgG4-RD mimickers fulfilled the corresponding diagnostic criteria.

Exclusion Criteria:

* Patients in pregnancy or preparing to pregnancy, patients with active infection, including HIV, HCV, HBV, TB, et al.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 300 IgG4-RD patients, 200 other autoimmune diseases, 60 IgG4-RD mimickers (pancreatic cancer, cholangiocarcinoma, vasculitis, lymphoproliferative diseases, inflammatory bowel disease, kimura disease) and 100 healthy controls were enrolled.
Sampling Method: Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-09-10 (Estimated)

PRIMARY OUTCOMES:
plasmablast/plasma cells in the diagnosis of IgG4-RD | 24 months
  plasmablast/plasma cells will be detected in IgG4-RD, other autoimmune disease and IgG4-RD mimickers at baseline.
plasmablast/plasma cells in relapse prediction of IgG4-RD | 24 months
  IgG4-RD patients will be followed up for at least 6 months. plasmablast/plasma cells will be detected at baseline, disease remission and disease relapse.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lin W, Zhang P, Chen H, Chen Y, Yang H, Zheng W, Zhang X, Zhang F, Zhang W, Lipsky PE. Circulating plasmablasts/plasma cells: a potential biomarker for IgG4-related disease. Arthritis Res Ther. 2017 Feb 10;19(1):25. doi: 10.1186/s13075-017-1231-2. PMID 28183334